CLINICAL TRIAL: NCT06785415
Title: Phase 1/2 Trial of Elotuzumab, Daratumumab, Iberdomide, and Dexamethasone for Relapsed Multiple Myeloma
Brief Title: Elotuzumab, Daratumumab, Iberdomide, and Dexamethasone for the Treatment of Relapsed Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC230812; NCI-2025-00138 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-010000 (Other: Mayo Clinic Institutional Review Board); MC230812 (Other: Mayo Clinic)
Record Dates: First submitted 2025-01-16; First posted 2025-01-21 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Biopsy; X-Rays; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; elotuzumab; iberdomide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (iberdomide, daratumumab, elotuzumab, dexamethasone) (Experimental): Patients receive iberdomide PO QD on days 1-21 of each cycle, daratumumab SC on days 1, 8, 15, 22 of cycles 1 and 2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles. Patients also receive elotuzumab IV on days 1, 8, 15, and 22 of cycles 1 and 2, and on day 1 of subsequent cycles and dexamethasone PO on days 1, 8, 15, and 22 of cycles 1-12 or at the discretion of the treating physician. Cycles repeat every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy during screening, on study and optionally at disease progression and CT, bone scan, MRI or PET/CT during screening, on study or at the discretion of the treating physician and EOT. Patients may undergo chest x-ray during screening.
  Interventions: Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Bone Scan; Procedure: Chest Radiography; Procedure: Computed Tomography; Biological: Daratumumab; Drug: Dexamethasone; Biological: Elotuzumab; Drug: Iberdomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
Procedure: Computed Tomography — Undergo CT and/or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Daratumumab — Given SC
  Other Names: Daratumumab Biosimilar HLX15; Daratumumab-fihj; Darzalex; HLX15; HuMax-CD38; JNJ 54767414; JNJ-54767414; JNJ54767414
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Biological: Elotuzumab — Given IV
  Other Names: BMS 901608; BMS-901608; BMS901608; Empliciti; HuLuc-63; HuLuc63; PDL 063; PDL-063; PDL063
Drug: Iberdomide — Given PO
  Other Names: CC 220; CC-220
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase I/II trial tests the safety, side effects, and best dose of iberdomide and how well it works in combination with daratumumab, elotuzumab, and dexamethasone in treating patients with multiple myeloma that has come back after a period of improvement (relapsed). Immunotherapy with iberdomide, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Daratumumab is in a class of medications called monoclonal antibodies. It binds to a protein called CD38, which is found on some types of immune cells and cancer cells, including myeloma cells. Daratumumab may block CD38 and help the immune system kill cancer cells. Elotuzumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Dexamethasone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Giving iberdomide in combination with daratumumab, elotuzumab, and dexamethasone may be safe, tolerable and/or effective in patients with relapsed multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the maximum tolerated dose (MTD) of the combination of iberdomide, daratumumab, elotuzumab, and dexamethasone (IberDEd) in patients with relapsed multiple myeloma (MM). (Phase 1 [Dose Confirmation Cohort]) II. To determine the proportion of patients with very good partial response (VGPR) or better with iberdomide, daratumumab, elotuzumab and dexamethasone (IberDEd) when used as therapy in patients with relapsed multiple myeloma. (Phase 2)

SECONDARY OBJECTIVES:

I. To assess the overall response rate (ORR) and complete response (CR or stringent complete response [sCR]) rate with the combination of iberdomide, daratumumab, elotuzumab and dexamethasone. (Phase 2) II. To assess the progression free survival and overall survival among patients with relapsed multiple myeloma following treatment with the combination of iberdomide, daratumumab, elotuzumab and dexamethasone. (Phase 2) III. To assess the time to response (defined as the time between the date of first dose and the first documented evidence of a partial response or better) following treatment with the combination of iberdomide, daratumumab, elotuzumab and dexamethasone in patients with relapsed MM. (Phase 2) IV. To describe the toxicities associated with the combination of iberdomide, daratumumab, elotuzumab and dexamethasone in patients with relapsed MM. (Phase 2)

CORRELATIVE RESEARCH:

I. Examine the proportion of next generation flow cytometry assessed minimal residual disease (MRD) negative complete response following therapy with iberdomide in combination with daratumumab, elotuzumab and dexamethasone. (Phase 2)

OUTLINE: This is a dose-escalation study of iberdomide followed by a dose-expansion study.

Patients receive iberdomide orally (PO) once daily (QD) on days 1-21 of each cycle, daratumumab subcutaneously (SC) on days 1, 8, 15, 22 of cycles 1 and 2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles. Patients also receive elotuzumab intravenously (IV) on days 1, 8, 15, and 22 of cycles 1 and 2, and on day 1 of subsequent cycles and dexamethasone PO on days 1, 8, 15, and 22 of cycles 1-12 or at the discretion of the treating physician. Cycles repeat every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy during screening, on study and optionally at disease progression and computed tomography (CT), bone scan, magnetic resonance imaging (MRI) or positron emission tomography (PET)/CT during screening, on study or at the discretion of the treating physician and end of treatment (EOT). Patients may undergo chest x-ray during screening.

After completion of study treatment, patients are followed up at 7 days then 30 days and every 3-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of signing the informed consent form (ICF).
* Diagnosis of relapsed multiple myeloma with ≤ 3 prior lines of therapy including treatment with proteasome inhibitors (i.e., ixazomib, carfilzomib, bortezomib), immunomodulatory imide drugs (i.e., lenalidomide, pomalidomide), and anti-CD38 drugs (i.e., daratumumab, isatuximab). Patients are required to have received a proteasome inhibitor, immunomodulatory imide drug, or combination of the two drug classes during first-line treatment.

  * Note: Prior treatment with iberdomide is not allowed. Patients should not be refractory simultaneously to all other drugs in the combination.
* Measurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2.
* Hemoglobin ≥ 8.0 g/dL (obtained ≤14 days prior to registration).
* Absolute neutrophil count (ANC) ≥ 1000/m^3 (obtained ≤14 days prior to registration).
* Platelet count ≥ 50,000/mm^3. Note: It is not permissible to transfuse subjects to achieve minimum platelet counts (obtained ≤14 days prior to registration).
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (≤ 3 x ULN for patients with Gilbert's syndrome) (obtained ≤14 days prior to registration).
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 2 x ULN and alkaline phosphatase ≤ 1.5 x ULN (obtained ≤14 days prior to registration).
* Calculated creatinine clearance ≥ 30 ml/min using the Cockcroft-Gault (obtained ≤14 days prior to registration).
* Negative pregnancy test done ≤ 7 days prior to registration, for persons of childbearing potential only. Note: A person of childbearing potential (PCBP) is a person who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months) and must:

  * Have 2 negative pregnancy tests prior to starting study treatment and must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.

AND

* Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with two forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting investigational product, during the study treatment, and for at least 28 days after the last dose of iberdomide, 90 days after the last dose of daratumumab, 7 months after last dose of elotuzumab whichever is longer.
* NOTE: Non-childbearing potential is defined as follows (by other than medical reasons):

  * ≥ 45 years of age and has not had menses for > 24 months.
  * Patients who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation.
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.

    * Willingness to follow Pregnancy Prevention Program requirements:
* Persons of childbearing potential must agree to use a contraceptive method that is highly effective (with a failure rate of < 1% per year), preferably with low user dependency, during the intervention period and for at least 7 months after the last dose of study intervention. These patients must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period.
* Persons able to father a child must agree that during the treatment intervention period and for 6 months after the last dose of study treatment (to allow for clearance of any altered sperm), the participant will:

  * Refrain from donating sperm while on study treatment, during dose interruptions and for at least 6 months following last dose of study treatment, PLUS either:
  * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, OR,
  * Must agree to use contraception/barrier such as a male condom (even if they have undergone successful vasectomy), and when having sexual intercourse with a person of childbearing potential who is not currently pregnant his partner will use an additional highly effective contraceptive method with a failure rate of < 1% per year.

    * Provide written informed consent.
    * Willingness to provide mandatory bone marrow specimens for correlative research.
    * Willing and able to adhere to the study visit schedule and other protocol requirements. Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
    * Willing to refrain from donating blood while on study treatment, during dose interruptions and for at least 28 days following the last dose of study treatment.

Exclusion Criteria:

* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Men or women of childbearing potential who are unwilling to employ adequate contraception.
* Receiving any other concurrent chemotherapy, or any ancillary therapy considered investigational.

  * Note: Bisphosphonates are supportive care rather than therapy and are thus allowed while on protocol treatment.
* Known to be human immunodeficiency virus (HIV) positive known or suspected active hepatitis C infection or seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]) at registration or ≤ 3 months prior to registration.

  * Note: Participants with resolved hepatitis B infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded.
  * EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
* Evidence of cardiovascular disease risk, as defined by any of the following:

  * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant electrocardiogram (ECG) abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block
  * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting ≤ three (3) months prior to registration.
  * Class III or IV heart failure as defined by the New York Heart Association functional classification system [NYHA, 1994]
  * Uncontrolled hypertension
  * History of life-threatening ventricular arrhythmias.
* Known moderate or severe persistent asthma, or currently has uncontrolled asthma of any classification.
* Unable or unwilling to undergo protocol required thromboembolism prophylaxis.
* Has taken a strong inhibitor or inducer of CYP3A4/5 including grapefruit, St. John's Wort or related products ≤ 14 days prior to registration.
* Known allergy to any of the study medications, their analogues or excipients in the various formulations.
* Major surgery ≤ 14 days prior to registration.
* Has been treated with an investigational agent (i.e., an agent not commercially available) ≤ 28 days or 5 half-lives (whichever is longer) prior to registration.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Any co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease.
* History of anaphylaxis or hypersensitivity to thalidomide, lenalidomide, or pomalidomide.
* Peripheral neuropathy grade ≥ 2.
* Severe acute respiratory syndrome coronavirus 2 infection ≤ 14 days prior to registration for mild or asymptomatic infections OR ≤ 28 days prior to registration for severe/critical illness.
* Gastrointestinal disease that may significantly alter the absorption of iberdomide.
* Received a live vaccine ≤ 90 days prior to registration.
* Prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years with the exception of the following noninvasive malignancies:

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin in situ (stage 0)
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is curative.
* Received hydroxychloroquine, quinacrine, chloroquine, methotrexate, leflunomide, sulfasalazine, mycophenolate mofetil, mycophenolic acid ≤ 28 days prior to registration.
* Received daily nonsteroidal anti-inflammatory drugs (NSAIDs) ≤ 14 days prior to registration. Note: Allowed if dose has been stable for at least 14 days.
* Received immunomodulating or immunosuppressive therapy as follows:

  * Etanercept ≤ 28 days prior to registration
  * Belimumab ≤ 12 weeks prior to registration
  * B-cell depleting or modulating agents (such as rituximab or anti-CD22 therapy) ≤ 365 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2031-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (Phase 1) | Up to 28 days
  The maximum tolerated dose (MTD) of the combination of iberdomide, daratumumab, elotuzumab, and dexamethasone (IberDEd) will be defined as the highest tested dose level that is determined to have acceptable toxicity and tolerability based on dose limiting toxicity definitions.
Proportion of patients with very good partial response (VGPR) or better (Phase 2) | Up to 3 years
  Will be defined as a patient who has achieved a VGPR, complete response (CR), or stringent complete response (sCR) and maintained it on two consecutive evaluations at any time during therapy per International Myeloma Working Group (IMWG) criteria.

SECONDARY OUTCOMES:
Overall response rate (Phase 2) | Up to 3 years
  Will be assessed as stringent Complete Response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), Minimal Response (MR), stable disease (SD), or progressive disease (PD).
Complete response rate (Phase 2) | Up to 3 years
  Will be estimated by the total number of patients who achieve sCR or CR.
Progression-free survival (Phase 2) | Up to 3 years
  Defined as the time from registration to the earliest date of documentation of disease progression, relapse, or death due to any cause.
Overall survival (Phase 2) | Up to 3 years
  Overall survival (OS) is defined as the time from registration to death due to any cause.
Time to response (Phase 2) | Up to 3 years
  Defined in patients who have achieved a response (PR or better) as the time from registration to the first incidence of a response.
Incidence of adverse events (AEs) (Phase 2) | Up to 3 years
  Will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The maximum grade for each type of AE will be recorded for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Binder, MD, MPH, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials